CLINICAL TRIAL: NCT07062523
Title: Application of [68Ga]Ga-FAPI-04 PET/CT in the Assessment of Inflammatory Activity in Sjögren's Syndrome
Brief Title: Analyse of Inflammatory Activity of Sjögren's Syndrome on 68Ga-FAPI PET-CT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-FAPI-pSS
Record Dates: First submitted 2024-06-28; First posted 2025-07-14 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-05

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-FAPI PET/CT in Sjögren's Syndrome (Experimental): All patients diagnosed with Sjögren's syndrome underwent 68Ga-FAPI PET/CT.
  Interventions: Drug: 68Ga-FAPI
- 68Ga-FAPI PET/CT in tumor patients (Experimental): Patients with tumors such as lung cancer and breast cancer, who had been excluded for Sjögren's syndrome, underwent 68Ga-FAPI PET/CT.
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 18.5-22.2MBq (0.5-0.6 mCi)/Kg 68Ga-FAPI. Tracer doses of 68Ga- FAPI will be used to image lesions of Sjögren's syndrome by PET/ CT.
  Other Names: 68Ga-Fibroblast activation protein Inhibitor

SUMMARY:
Sjögren's syndrome (SS) is a chronic autoimmune disease primarily affecting the salivary and lacrimal glands, leading to symptoms of dryness. Assessing the inflammatory activity is crucial for guiding treatment. Fibroblast activation protein (FAPI) PET is an emerging imaging technique increasingly used for evaluating various inflammations and tumors. Thus this prospective study is going to investigate the uptake characteristics of FAPI PET in Sjögren's syndrome and evaluate its potential in assessing inflammatory activity to guide clinical treatment. A control group of tumor patients undergoing FAPI PET imaging will be included to compare FAPI uptake patterns between autoimmune inflammation and neoplasia.

DETAILED DESCRIPTION:
Sjögren's syndrome (SS), characterized by its chronic autoimmune nature, predominantly targets the salivary and lacrimal glands, resulting in the classic symptoms of dry mouth and dry eyes. This condition can extend beyond these glands, impacting other systems in the body and leading to a variety of clinical manifestations, such as fatigue, joint pain, and in more severe cases, an increased risk of lymphoma. The heterogeneity of SS, with its potential to affect multiple organs, underscores the importance of accurately assessing the level of inflammation when developing a treatment plan.

Fibroblast activation protein (FAPI) PET imaging is a cutting-edge diagnostic tool that has shown promise in the detection and evaluation of inflammation associated with a range of pathologies, including various tumors. This innovative imaging technique takes advantage of the elevated levels of FAPI, a protein that is overexpressed in cancer-associated fibroblasts, which are a common feature in numerous malignant solid tumors. Moreover, FAPI's role in inflammation suggests its potential as a biomarker for disease activity in conditions like SS.

The prospective study mentioned aims to delve deeper into the utility of FAPI PET in the context of SS. It will explore how FAPI PET imaging can be applied to visualize and quantify inflammatory changes within the salivary and lacrimal glands, which are typically affected in SS. The study will involve a cohort of SS patients who will undergo FAPI PET scans, and the findings will be correlated with their clinical symptoms, serological markers of inflammation, and other imaging modalities.

The primary objective of this study is to determine the uptake characteristics of FAPI PET in patients with SS, providing valuable data on the distribution and intensity of FAPI uptake in affected tissues. By analyzing these patterns, researchers can assess whether FAPI PET imaging can serve as a reliable and sensitive biomarker for inflammatory activity in SS. This information could be instrumental in guiding clinical treatment decisions, predicting treatment responses, and identifying potential disease flares.

If the study confirms the effectiveness of FAPI PET in assessing inflammation in SS, it could revolutionize the way the disease is monitored and managed. The ability to non-invasively visualize and quantify inflammation could lead to more personalized treatment strategies, more precise disease monitoring, and ultimately, improved outcomes for individuals living with SS. Furthermore, this research could also open up new avenues for understanding the pathophysiology of SS and other autoimmune conditions, potentially leading to the development of novel therapeutic targets and approaches.

The study will also include a control group of patients with various tumors who are scheduled for 68Ga-FAPI PET/CT as part of their diagnostic workup. This will allow for a comparative analysis of FAPI uptake between inflammatory and malignant lesions, enhancing the specificity assessment of FAPI PET in autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Fulfillment of the 2016 ACR-EULAR Classification Criteria for pSS at enrollment. OR diagnosis of a solid tumor scheduled for FAPI PET imaging

Exclusion Criteria:

* Combined with tumors or other connective tissue diseases (for SS group);
* Patients who are currently using hormones/biological agents (for both groups)；
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Optimal imaging time | up to 3 month
  Patients were included for PET dynamic imaging to find the optimal imaging time for FAPI PET in Sjögren's syndrome
Correlation with inflammatory markers | 6 weeks
  Inflammatory and immune markers (e.g., IL-6, TNF-α, CRP) were measured using enzyme-linked immunosorbent assay (ELISA) in all patients, and correlational analysis was performed with PET uptake values.
Comparative uptake analysis between Sjögren's syndrome and tumor patients | up to 3 months
  Comparison of standardized uptake values (SUV) and distribution patterns of 68Ga-FAPI in salivary/lacrimal glands of SS patients versus tumor lesions in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT07062523/Prot_SAP_ICF_000.pdf